CLINICAL TRIAL: NCT07317401
Title: REenergizeME: Oxygen Therapy (OT) as a Novel Treatment for Post-Viral Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Brief Title: Investigating the Effects of Intermittent Hypoxia-Hyperoxia Treatment (IHHT) in People With Post-Viral Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) to Improve Fatigue, Pain, and Quality of Life by Targeting Mitochondrial Dysfunction and Autonomic Nervous System Impairment
Acronym: REenergizeME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sagsnr.: 2500959; 10.46540/3165-00221B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) (ICD-10 G93.3)
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent hypoxia-hyperoxia treatment (IHHT) (Active Comparator): An individualized treatment is administered to patients in 4-7 intervals, within 22-40 minutes. Blood oxygen saturation (O2-Sat) rises and falls cyclically, due to fluctuating fractions of inspired oxygen (FiO2): 9-13% in the hypoxic phase and 36% in the hyperoxic restitution phase.
  Interventions: Other: Intermittent hypoxia-hyperoxia treatment (IHHT)
- Sham treatment (Placebo Comparator): The placebo group will undergo 'sham treatment' with air breathing at 21% FiO2. To equate the sensation of IHHT, airbrakes will be simulated similar to the IHHT intervals in the treatment protocol.
  Interventions: Device: Placebo

INTERVENTIONS:
Other: Intermittent hypoxia-hyperoxia treatment (IHHT) — The apparatus used to deliver the IHHT is the CellOxy machine (TUR GmbH, Rostock, Germany, CE Medical device class IIa). The CellOxy machine is constructed with a built-in compressor, an air reservoir, and a set of membranes, making it possible for the machine to either add or remove oxygen from the atmospheric air, thus delivering a dynamic FiO2 (fraction of inspired oxygen). The individualized therapy settings are regulated via the attached user interface. It is connected to a desk monitor and a data-collecting server.
  Arms: Intermittent hypoxia-hyperoxia treatment (IHHT)
Device: Placebo — The placebo group will undergo 'sham treatment' with air breathing at 21% FiO2. To equate the sensation of oxygen therapy, airbrakes will be simulated similar to the oxygen therapy intervals in the treatment protocol.
  Arms: Sham treatment

SUMMARY:
This study is testing a new treatment for people with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) and long-term symptoms after COVID-19. Both conditions cause extreme fatigue, muscle pain, "brain fog," and trouble concentrating, which often get worse after physical or mental activity. Currently, no effective treatments are available.

The treatment being studied is called Intermittent Hypoxia-Hyperoxia Treatment (IHHT). It uses a machine called CellOxy to deliver short cycles of low oxygen (hypoxia) and high oxygen (hyperoxia) through a mask. Each session lasts 22-40 minutes and is carefully monitored to track oxygen levels, heart rate, and breathing. The therapy is customized for each patient to ensure comfort and effectiveness. IHHT is believed to help the body adapt to oxygen-related stress, improving energy production and reducing inflammation.

In this trial, 87 patients with ME/CFS will be randomly assigned to receive either IHHT or a placebo treatment with normal oxygen levels over six weeks. The placebo group will follow a similar procedure without oxygen changes. An additional 17 healthy individuals will be recruited as a comparison group, but they will not undergo the treatment.

Participants will have medical check-ups before and after treatment to evaluate changes in fatigue, mental sharpness, pain, autonomic nervous system function, and overall quality of life. Blood samples and small skin biopsies will also be taken to study the biological processes behind ME/CFS and how the treatment works.

This research aims to find out if IHHT can improve the lives of people with ME/CFS or long-term COVID symptoms. The results could also provide new insights into the causes of these challenging conditions and guide future treatments.

ELIGIBILITY:
Eligibility Criteria ME/CFS Patients

Inclusion Criteria:

* Established diagnosis of ME/CFS according to the International Consensus Criteria (ICC)
* Presence of post-exertional malaise (PEM)
* Disease duration > 6 months
* Mild or moderate disease severity according to NICE guidelines
* Ability to attend clinic visits for inclusion and IHHT intervention
* Female sex
* Age 20-59 years

Exclusion Criteria:

* Not meeting the International Consensus Criteria for ME/CFS
* Disease severity classified as severe according to NICE guidelines
* Inability to attend clinic visits
* Male sex
* Age < 20 or > 59 years

Healthy Controls

Inclusion Criteria:

* Ability to attend clinic visits
* Female sex
* Age 20-59 years
* BMI matched to ME/CFS participants
* Activity level matched to ME/CFS participants

Exclusion Criteria:

* History or current diagnosis of ME/CFS
* Inability to attend clinic visits
* Male sex
* Age < 20 or > 59 years

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in quality of life vitality score (energy level and fatigue) using the self-reported SF-36 questionnaire. | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No